CLINICAL TRIAL: NCT01411540
Title: Effects of Diet on Body Composition
Brief Title: Effects of a Wholegrain Diet on Body Composition and Energy Balance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Principal Investigator, John Kirwan, Staff, Department of Pathobiology, The Cleveland Clinic
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 10-434
Record Dates: First submitted 2011-07-27; First posted 2011-08-08 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Overweight; Obesity; Pre-diabetic
Keywords: Body composition; Health markers; Diet
MeSH Terms: conditions — Overweight; Obesity; Glucose Intolerance | interventions — Whole Grains; Diet; Body Composition

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Whole grain diet (Experimental): Subjects will eat a whole grain based diet for eight weeks. Pre-and post-diet intervention testing will determine effects on body composition. Whole grain-based are will be compared to the refined grain based diet.
  Interventions: Dietary Supplement: Whole grains
- Refined grain diet (Active Comparator): Subjects will eat a refined grain diet for 8 weeks matched with the whole grain arm for calorie and macro nutrient intake. Pre-and post-diet testing will determine effects on body composition.
  Interventions: Dietary Supplement: Whole grains

INTERVENTIONS:
Dietary Supplement: Whole grains — Comparison of a diet containing whole grain compared to an energy matched diet based on similar foods, but using refined grains.
  Other Names: Diet; Body composition

SUMMARY:
The purpose of this study is to compare a diet containing whole grains versus an energy matched diet using refined grains on body composition and metabolism.

DETAILED DESCRIPTION:
The investigators hypothesis is that a diet high in whole-grains reduces abdominal fat. These findings might have clinical and public health significance for reducing obesity and related co-morbidities like type 2 diabetes and cardiovascular disease. Using a double-blind cross-over design, energy expenditure, body composition and metabolic health will be assessed. Three day inpatient study visits to the Cleveland Clinic Clinical Research Unit (CRU) will be implemented for metabolic control and testing. Total daily energy expenditure will be measured using the doubly labeled water (DLW) method. Body fat and glucose/protein metabolism will be assessed by imaging and isotope techniques, respectively. Blood, urine, and stool samples will also be collected for cardiometabolic and digestive health outcomes. After baseline testing, subjects will begin an 8 week dietary intervention, where all food and non-water beverages will be supplied by the study center. Dietary compliance will be assessed by weigh back measurements two times a week. To assess time course effects of diets differing in the amount of fiber on body composition and metabolic health, subjects will provide plasma and urine samples 2, 4, and 8 weeks after initial testing. Imaging and isotope analysis will be performed baseline and at week 8. All post testing will be conducted after week 8 following similar pre-testing control conditions. Subjects will then undergo an 8-10 week washout period where they will be instructed to return to their normal diet (except for any supplements). After the washout period, subjects will start the second arm of the intervention and consume the alternate diet (i.e. refined or whole grain diet). All energy expenditure, body composition and metabolic testing procedures will be repeated during the alternative arm of the study as described above.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 20-50 years
* BMI between 25 and 38 kg/m2
* Normal whole grain intake <1 serving/d (Appendix 1)
* Low average consumption of alcohol (<1 standard drink/day; <7 standard drinks/week)
* Non-smoker
* No major chronic illness
* Fasting glucose <126 mg/dl
* Able to access the study centre (Lerner Research Institute and the Clinical Research Unit at the Cleveland Clinic) throughout the study
* Have access to a microwave oven and refrigerator/freezer

Exclusion Criteria:

* Any known food allergy with the possibility to result in a serious adverse reaction, or an allergy to a food item that cannot be removed from the diet (i.e. peanuts).
* Aversion or dislike to study foods
* Regular use of dietary supplements and not willing/able to stop usage during the study period
* Cardiovascular conditions including significant known coronary artery disease, arrhythmia, known peripheral vascular disease (large vessel disease), uncompensated congestive heart failure, history of stroke, or uncontrolled hypertension (defined as medically treated with the mean of 3 separate measurements SBP > 180 mm Hg or DBP > 110 mm Hg)
* Severe pulmonary disease defined as FEV1 < 50% of predicted value
* Kidney disease including diagnosed chronic kidney disease, renovascular hypertension, renal artery stenosis, or chronic renal insufficiency with a creatinine level > 1.8 mg/dl
* Known history of chronic liver disease (except for NAFLD), hepatitis, positive serologic test result for hepatitis B surface antigen and/or hepatitis C antibody, α-1-antitrypsin deficiency
* GI disorders including a known history of celiac disease and/or any other malabsorptive disorders or inflammatory bowel disease (Crohn's disease or ulcerative colitis)
* Psychiatric disorders including dementia, active psychosis, severe depression (requiring > 2 medications), history of suicide attempts, alcohol or drug abuse within the previous 12 months
* Other known metabolic disease such as clinical hypothyroidism and hyper thyroidism, Graves Disease, thyroid cancer, nodules or multinodular goiter
* Malignancy within five years (except squamous cell and basal cell cancer of the skin)

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2010-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in body composition | 24 months
  The primary outcome is the change in body composition after an eight-week intervention of either whole grains or refined grains, corrected for baseline body composition at the start of the appropriate treatment arm.

SECONDARY OUTCOMES:
Total energy expenditure | Eight-week cross-over trial with 10 week washout period between intervention arms.
  DLW will be used to assess total daily energy expenditure (TDEE).
Glucose turnover | Eight weeks
  Glucose turnover will be assessed by [U-13C] glucose and [6,6-(2)H] glucose kinetics from breath, plasma and urine samples.
Protein turnover | Eight weeks
  Protein turnover will be examined using 13C-leucine and 15N-glycine kinetics in breath, plamsa, and urine samples.

CONTACTS AND LOCATIONS:
Overall Officials: John P. Kirwan, Ph.D., Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Mey JT, Godin JP, Scelsi AR, Kullman EL, Malin SK, Yang S, Floyd ZE, Poulev A, Fielding RA, Ross AB, Kirwan JP. A Whole-Grain Diet Increases Whole-Body Protein Balance Compared with a Macronutrient-Matched Refined-Grain Diet. Curr Dev Nutr. 2021 Sep 25;5(11):nzab121. doi: 10.1093/cdn/nzab121. eCollection 2021 Nov. PMID 34805723
- [Derived] Malin SK, Kullman EL, Scelsi AR, Haus JM, Filion J, Pagadala MR, Godin JP, Kochhar S, Ross AB, Kirwan JP. A whole-grain diet reduces peripheral insulin resistance and improves glucose kinetics in obese adults: A randomized-controlled trial. Metabolism. 2018 May;82:111-117. doi: 10.1016/j.metabol.2017.12.011. Epub 2018 Jan 3. PMID 29305946
- [Derived] Kirwan JP, Malin SK, Scelsi AR, Kullman EL, Navaneethan SD, Pagadala MR, Haus JM, Filion J, Godin JP, Kochhar S, Ross AB. A Whole-Grain Diet Reduces Cardiovascular Risk Factors in Overweight and Obese Adults: A Randomized Controlled Trial. J Nutr. 2016 Nov;146(11):2244-2251. doi: 10.3945/jn.116.230508. Epub 2016 Oct 19. PMID 27798329